

## DATA ANALYSIS PLAN

Analysis will be on an intention-to-treat basis. Outcomes will be analyzed at two time-points (12 and 24 weeks). Analysis of covariance will be used to test for differences in weight loss between groups at each time point. The models will be fitted using linear regression with weight as the outcome variable, treatment group as the predictor variable of interest and weight at baseline included as a covariate. Age, gender, dietary intake (kilocalories) and physical activity at baseline will enter the model for adjustment. Statistical significance of the primary efficacy analysis (at 12 and 24 weeks) will be based on Hochberg's multiple testing procedure with the family wise error rate for each time point held at 2.5%. Secondary hypothesis tests will be performed using a 2-sided 5% significance level.